CLINICAL TRIAL: NCT06463132
Title: Phase 1b Open-Label, Multi-Center, Randomized Trial to Evaluate the Safety of PEP and EUFLEXXA for the Treatment of Subjects With Knee Osteoarthritis (KOA)
Brief Title: Phase 1b Clinical Trial to Evaluate PEP and EUFLEXXA for Knee Osteoarthritis (KOA)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rion Inc. (Industry)
Collaborators: Caidya Clinical Research Organization (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO-00126
Record Dates: First submitted 2024-06-07; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Exosome; Osteoarthritis; Joint Disease; Hyaluronic Acid; Extracellular Vesicle; Musculoskeletal Diseases; Arthritis; Randomized Clinical Trial; Rheumatic Diseases; Osteoarthritis, Knee; Biologic
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Joint Diseases; Musculoskeletal Diseases; Arthritis; Rheumatic Diseases

STUDY DESIGN:
Intervention Model Description: Arm 1A, PEP Low Dose Arm 1B, PEP High Dose Arm 2A, PEP-EUFLEXXA Low Dose Arm 2B, PEP-EUFLEXXA High Dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- 1A PEP Low Dose (Experimental): 1A PEP Low Dose in Saline
  Interventions: Drug: PEP
- 1B PEP High Dose (Experimental): 1B PEP High Dose in Saline
  Interventions: Drug: PEP
- 2a PEP-EUFLEXXA Low Dose (Experimental): 2A PEP-EUFLEXXA Low Dose
  Interventions: Combination Product: PEP/Euflexxa
- 2b PEP-EUFLEXXA High Dose (Experimental): 2B PEP-EUFLEXXA High Dose
  Interventions: Combination Product: PEP/Euflexxa

INTERVENTIONS:
Combination Product: PEP/Euflexxa — Euflexxa (PMA: P010029)
  Arms: 2a PEP-EUFLEXXA Low Dose; 2b PEP-EUFLEXXA High Dose
Drug: PEP — PEP (Purified Exosome Product)
  Arms: 1A PEP Low Dose; 1B PEP High Dose

SUMMARY:
Evaluate the safety and exploratory efficacy of single intra-articular injections of PEP reconstituted with 0.9% Normal Saline at a low dose (one vial PEP) and high dose (two vials PEP), with and without EUFLEXXA, for the treatment of Knee Osteoarthritis

DETAILED DESCRIPTION:
Study Plan (with Dose Escalation): Arm 1 and Arm 2 will run in parallel such that initially 3 subjects will be enrolled in Arm 1a (PEP Low Dose) and 3 subjects will be enrolled in Arm 2a (PEP-EUFLEXXA Low Dose). After all 6 subjects complete the 30 day follow up and there was not more than 1 AE grade 3 or higher per Arm, a further 9 subjects will be enrolled in Arm 1b (PEP High Dose) and a further 9 subjects will be enrolled in Arm 2b (PEP-EUFLEXXA High Dose).

ELIGIBILITY:
Inclusion Criteria:

• Age: Adults aged 18-90 years of age

Type of Participant and Disease Characteristics:

* Diagnosis of unilateral or bilateral symptomatic KOA of at least 6 months duration (meets American College of Rheumatology/Arthritis [ACR] criteria)
* Daily knee pain in the more symptomatic knee of ≥ 30 and ≤ 80 on a 100-point VAS for greater than 6 months
* Kellgren Lawrence Grade 2 to 3 osteoarthritis in the more symptomatic knee based on standard knee radiographs
* Failed conservative management including at least 2 of the following:
* Lack of improvement with attempted weight loss in the past year if body mass index (BMI) > 30 kg/m2;
* Lack of response to a 4-week trial in the past year of oral acetaminophen or NSAIDs taken as needed;
* Lack of response to a 4-week trial in the past year of topical NSAIDs or capsaicin applied as needed;
* Lack of improvement after injection therapy with cortisone, PRP or hyaluronic acid;
* Lack of improvement after a 4-week course of physical therapy in the past year; or
* Lack of improvement after a 4-week trial of quadriceps strengthening home exercise program in the past year.
* Requesting injection therapy for pain management
* Contraceptive use by participants and their partners should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  o A serum pregnancy test (human chorionic gonadotropin [hCG]) should be done for all women of childbearing potential (WOCBP) at Screening, and a urine pregnancy test should be done on Day 1, prior to injection, with results reviewed before injection to confirm the participant's eligibility. Participants who have positive pregnancy test result will not be permitted to continue in the study (see Section 5.2, Exclusion criteria 18 and 19).
* Signed informed consent as described in Appendix 1 (Section 10.1) which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Ability to comply with protocol.

Exclusion Criteria:

* Steroid or viscosupplement injection in the planned treatment knee(s) within the past 3 months.
* PRP injection in the planned treatment knee(s) within the past 6 months.
* History of documented allergy to intra-articular EUFLEXXA.
* History of cancer including melanoma (with the exception of localized skin cancer) in the past 2 years.
* HIV positive participants.
* BMI > 40 kg/m2.
* Arthroscopic debridement in the planned treatment knee(s) in the last 6 months.
* Cartilage restoration procedure in the planned treatment knee(s) in the last 5 years.
* History of gout or pseudogout.
* History of or evidence of active rheumatologic disease, severe peripheral neuropathy, clinically evident cardiac or respiratory disease that interferes with functional status.
* Poorly controlled diabetes defined as a glycated hemoglobin (HbA1c) concentration of ≥ 8.0%.
* Currently taking any cancer treatment regimen (including aromatase inhibitors).
* Calcium pyrophosphate deposition disease (CPPD) evident on X-ray.
* Systemic (oral, intravenous, or intramuscular) steroids in the last 3 months.
* Concurrent participation in another investigational drug or device study or participation in the last 30 days prior to enrollment.
* Evidence of recent alcohol or drug abuse, or history of medication misuse or addiction.
* Female participants who are pregnant, breast feeding, or trying to become pregnant.
* Women unwilling to use approved contraception method for 3 months after receiving dose of investigational drug.
* Unwilling or unable to comply with Telehealth visits (eg, ability to access internet, on camera capabilities, etc).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Follow up 90 Days post injection occurrence of DLTs | First 90 days
  The safety of a single intra-articular injection of PEP, with or without EUFLEXXA, through the initial 90-day treatment period as assessed by the occurrence of DLTs with severity grading based on the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI CTCAE).
Long Term Safety Follow-Up Occurrence of DLTs From Day 91 to Day 365 | Day 365
  The long-term safety after treatment with a single intra-articular injection of PEP, with or without EUFLEXXA as assessed from the incidence of DLTs during the Day 91 through Day 365 follow up period.

SECONDARY OUTCOMES:
Exploratory Endpoints of Efficacy-Radiographic Response | Day 365
  Radiographic response, evaluated pre- and post-injection by an independent, blinded radiologist's assessment:
  Decrease or lack of progression of cartilage damage (thickness, denudation) and/or bone marrow edema on magnetic resonance imaging (MRI) at 6 or 12 months after injection Decrease or lack of progression in joint space narrowing on weight bearing X ray at 12 months after injection
Exploratory Endpoints of Efficacy-Participant-Reported responses: | Day 365
  Clinical improvement measured using a 100 point pain visual analogue scale (VAS) and modified Western Ontario and McMasters University Arthritis Index Questionnaire (WOMAC), which utilizes measures of pain and function, and treatment success based on Osteoarthritis Research Society International Outcome Measures in Rheumatology (OARSI OMERACT) responder criteria defined as follows:
  Absolute change of 20 points or more on the VAS 100-point scale; or Improvement of 50% of more in the modified WOMAC pain or function score; or Absolute change of 20 points or more in the combined modified WOMAC pain and function score.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No